CLINICAL TRIAL: NCT03610074
Title: Relieve the Patient's Thirst, Refresh the Mouth First
Brief Title: Relieve the Patient's Thirst, Refresh the Mouth First (ICU-MIC)
Acronym: ICU-MIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Arras (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017-03
Record Dates: First submitted 2018-06-21; First posted 2018-08-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Hypernatremia; Dehydration
Keywords: thirst; mouth; critical care; water deprivation
MeSH Terms: conditions — Hypernatremia; Dehydration | interventions — Hematologic Tests

STUDY DESIGN:
Intervention Model Description: Adult patient displaying an hypernatremia upper than 150mmol/L or an hypernatremia upper than 145mmol/L associated with a water deficiency upper than 3L
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mint ice cubes (Experimental): Physician applies 3 mint ice cubes in mouth of highly dehydrated patient. Patient undergoes an additional blood test at 5 min from mint ice cubes application.
  Physician performs patient's questioning before mint ice cubes application and at 5 min, 1h, 2h, 4h, 12h and 24h from mint ice cubes application.
  Interventions: Other: Mint Ice Cube; Procedure: Blood test; Other: Patient's questioning

INTERVENTIONS:
Other: Mint Ice Cube — Application in patient's mouth of 3 mint ice cubes
Procedure: Blood test — Additional blood test 5 min after mint ice cubes application
Other: Patient's questioning — Patient's questioning before mint ice cubes application and at 5 min, 1h, 2h, 4h, 12h and 24h from mint ice cubes application

SUMMARY:
Thirst is considered as one of the most distressing symptoms experienced by patients hospitalized in the Intensive Care Unit (ICU). Whereas pain is a permanent concern for all caregivers, thirst is often ignored and its complications are poorly known. Mechanisms involved in thirst regulation are numerous and complex. To date, care of thirst is still non optimal. Critically ill patients are usually rehydrated intravenously or using a naso-gastric tube, thus shunting the mouth as a therapeutic target to relieve the patient's thirst.

Water, cold and mint applied in mouth were studied separately and were shown to decrease thirst significantly on animal models and healthy humans.

Therefore, the hypothesis of this study is that application of small mint ice cubes in mouth of very dehydrated ICU patients should allow decreasing quickly and significantly thirst for these patients, before the correction of their biological parameters, like natremia and osmolarity.

ELIGIBILITY:
Inclusion Criteria:

* Hypernatremia upper than 150mmol/L or hypernatremia upper than 145mmol/L associated with water deficiency upper than 3L
* Estimated hospitalization duration in ICU upper than 24h

Exclusion Criteria:

* Contraindication for ice cubes application in mouth
* Known mint allergy
* Incapability to understand study outcome and to answer basic questions
* Pregnancy
* Dying person

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-03-08 (Actual)

PRIMARY OUTCOMES:
Change of thirst intensity at 5 minutes from mint ice cubes application | at 5 minutes from mint ice cubes application
  The primary endpoint is a change of thirst intensity of at least 1.5 points on the thirst intensity scale at 5 minutes from mint ice cubes application. Thirst intensity scale is a numeric scale ranging from 0 to 10 points. 0 corresponds to no thirst (the best outcome). 10 corresponds to a thirst of the strongest possible intensity (the worst outcome).

SECONDARY OUTCOMES:
Change of thirst-associated discomfort at 5 minutes from mint ice cubes application | at 5 minutes from mint ice cubes application
  This secondary endpoint is a change of thirst-associated discomfort on the discomfort scale at 5 minutes from mint ice cubes application. The discomfort scale is a numeric scale ranging from on a 0 to 5 points. 0 corresponds to "very comfortable" (the best outcome). 5 corresponds to "very uncomfortable" (the worst outcome).
Time of appearance of the observed effect on thirst intensity | over 24 hours from mint ice cubes application
  This secondary endpoint is the delay (in minutes) between mint ice cubes application and the observed effect on thirst intensity.
Duration of the observed effect on thirst intensity | over 24 hours from mint ice cubes application
  This secondary endpoint measures how much time (in minutes) mint ice cubes application keeps working on thirst intensity.
Change of natremia at 5 minutes from mint ice cubes application | at 5 minutes from mint ice cubes application
  Natremia (in mmol/L)
Change of natremia at 24 hours from mint ice cubes application | at 24 hours from mint ice cubes application
  Natremia (in mmol/L)
Change of plasma osmolarity at 5 minutes from mint ice cubes application | at 5 minutes from mint ice cubes application
  Plasma osmolarity (in mmol/L)
Change of plasma osmolarity at 24 hours from mint ice cubes application | at 24 hours from mint ice cubes application
  Plasma osmolarity (in mmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm LEMYZE, MD, Principal Investigator — Centre Hospitalier Arras
Locations (2):
- France (2):
  - Centre Hospitalier d'Arras, Arras
  - Centre Hospitalier de Lens, Lens

IPD SHARING:
Plan to Share IPD: No